CLINICAL TRIAL: NCT05995808
Title: Cyclin D1 as a Prognostic Factor in Multiple Myeloma and Its Association With the Immunological Prognostic Factor PDL1 and Clinical and Biochemical Lab Tests
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Fainan Khaled Ahmed, clinical pathology specialist, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med-23-07-02MD
Record Dates: First submitted 2023-08-09; First posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- diagnostic group (Experimental)
  Interventions: Procedure: Bone marow biopsy and aspiration; Diagnostic Test: biochemical and heamatological tests

INTERVENTIONS:
Procedure: Bone marow biopsy and aspiration — Bone marrow biopsy and biopsy aspiration
Diagnostic Test: biochemical and heamatological tests — complete blood count ,serum urea and creatinine
  Other Names: complete blood count ,urea and creatinine in serum

SUMMARY:
Multiple myeloma (MM) is the most common bone marrow malignancy of terminally differentiated plasma cells. It accounts for about 1% of all malignant diseases and 10% of haematological malignancies and takes the second place after non-Hodgkin lymphoma .

There are some serological and clinical criteria that help to detect the stage of MM and predict the patients' prognosis. These criteria include the level of M protein, calcium, haemoglobin, albumin, creatinine, β2-microglobulin and glomerular filtration rate (GFR).

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 18 year with newly diagnosed MM.
2. Approval to sign an informed written consent.

Exclusion Criteria:

* 1. Patient younger than 18 years. 2.Refusal to sign an informed written consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Cycline D1 expression in bone marrow biopsy of multiple myeloma patient | 1 year
  Cycline D1 expression in bone marrow biopsy of multiple myeloma patient